CLINICAL TRIAL: NCT00823667
Title: Palliative Care for Quality of Life and Symptom Concerns in Early Stage Lung Cancer
Brief Title: Effects of Palliative Care on Quality of Life and Symptom Control in Patients With Stage I, Stage II, or Stage IIIA Non-Small Cell Lung Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08034; P01CA136396 (NIH); P30CA033572 (NIH); CHNMC-08034; CDR0000631255 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Early Intervention, Educational; Therapeutics; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1 Usual care (Active Comparator)
  Interventions: Other: medical chart review; Other: questionnaire administration; Procedure: end-of-life treatment/management; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment
- Phase 2 Intervention (Active Comparator)
  Interventions: Other: educational intervention; Other: medical chart review; Other: questionnaire administration; Procedure: end-of-life treatment/management; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: educational intervention — Palliative care intervention at weeks 3,4,5 and 6 post study enrollment
  Arms: Phase 2 Intervention
Other: medical chart review — Occurs at 1 year post study enrollment
Other: questionnaire administration — Occurs at baseline, 6 weeks, 12 weeks, 24 weeks, 36 weeks and 52 weeks post study enrollment
Procedure: end-of-life treatment/management — Occurs at baseline, 6 weeks, 12 weeks, 24 weeks, 36 weeks and 52 weeks post study enrollment
Procedure: psychosocial assessment and care — Occurs at baseline, 6 weeks, 12 weeks, 24 weeks, 36 weeks and 52 weeks post study enrollment
Procedure: quality-of-life assessment — Occurs at baseline, 6 weeks, 12 weeks, 24 weeks, 36 weeks and 52 weeks post study enrollment

SUMMARY:
RATIONALE: Palliative care may be more effective than standard care in improving quality of life and symptoms in patients with lung cancer.

PURPOSE: This clinical trial is studying the effects of palliative care on quality of life and symptom control in patients with stage I, stage II, or stage IIIA non-small cell lung cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the effects of palliative care intervention (PCI) vs standard care on overall quality of life and psychological distress in patients with resectable stage I-IIIA non-small cell lung cancer.
* To compare symptom control in these patients.
* To compare geriatric assessment outcomes, as measured by OARS (Older Americans Resources and Services) Instrumental Activities of Daily Living, MOS Activities of Daily Living, MOS (Medical Outcomes Study)Social Activities Limitation Scale, Hospital Anxiety and Depression Scale scores, and Karnofsky performance scale, in these patients.
* To compare the effects of the PCI vs standard care on resource use.
* To identify subgroups of patients who benefit most from the PCI in relation to sociodemographic characteristics, treatment factors, and geriatric assessment predictors at week 12.

OUTLINE: Patients assigned to 1 of 2 groups.

* Group I (standard care): Patients receive standard care. Patients complete questionnaires at baseline and at 6, 12, 24, 36, and 52 weeks to evaluate quality of life (QOL), symptoms, psychological distress, and geriatric assessments. A medical chart review is performed at 52 weeks to assess the progression of treatment, episodes of care, and re-admissions.
* Group II (palliative care intervention): Patients receive an individualized interdisciplinary palliative care intervention combining patient-centered teaching principles and concepts that are learner-centered (builds on the strengths, interests, and needs of the learner), knowledge-centered (teacher is proficient in the content being taught), assessment-centered (learners are given an opportunity to test their understanding and receive feedback), and community-centered (opportunities are available for continued learning and support). Patients undergo 4 teaching sessions (based on the patient-centered teaching principles and concepts) that focus on physical, psychological, social, and spiritual well-being, respectively, once a week in weeks 3-6. Patients then receive 4 follow-up phone calls in weeks 9-21 to clarify questions or review concerns from the teaching sessions and to coordinate follow-up resources as needed. Patients also complete questionnaires as in group I.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I-IIIA resectable NSCLC - Undergoing either lobectomy, pneumonectomy, segmentectomy, or wedge resection
* Living within a 50 mile radius of the City of Hope
* No previous cancer within the past 5 years

Exclusion Criteria:

* Diagnosis of stage II-III NSCLC that are not resectable based on clinical and individual characteristics (co-morbidities, extent of disease, bulky mediastinal lymph nodes [N2], etc.)
* NSCLC patients receiving radiofrequency ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2009-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Overall quality of life and psychological distress | 1 year after study enrollment
Symptom control | 1 year after study enrollment
Geriatric assessment outcomes as measured by OARS Instrumental Activities of Daily Living, MOS Activities of Daily Living, MOS Social Activities Limitation Scale, Hospital Anxiety and Depression Scale scores, and Karnofsky performance scale | 1 year after study enrollment
Resource use as measured by chart audits | 1 year after study enrollment
Identification of subgroups of patients who benefit most from the palliative care intervention in relation to sociodemographic characteristics, treatment factors, and geriatric assessment predictors at week 12 | Week 12 after study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Betty Ferrell, PhD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States

REFERENCES:
- [Derived] Kim JY, Sun V, Raz DJ, Williams AC, Fujinami R, Reckamp K, Koczywas M, Cristea M, Hurria A, Ferrell B. The impact of lung cancer surgery on quality of life trajectories in patients and family caregivers. Lung Cancer. 2016 Nov;101:35-39. doi: 10.1016/j.lungcan.2016.08.011. Epub 2016 Aug 30. PMID 27794406